CLINICAL TRIAL: NCT06248580
Title: Find HDV and Determine Its Status in Turkey "SITU(HD)VATION"
Brief Title: Find HDV and Determine Its Status in Turkey
Acronym: SITUHDVATION
Status: Recruiting | Type: Observational
Sponsor: Yaşar Bayındır, MD (Other)
Collaborators: SOUTHEAST NEUROLOGY AND INFECTIOUS DISEASES SOCIETY (Unknown); Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Yaşar Bayındır, MD, Chief Physician, Prof. Dr., M.D., Guven Health Group
Organization: Guven Health Group (Other)
Other Study IDs: Guven Health Group
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Chronic Hepatitis D Infection; Fibrosis, Liver; Hepatocellular Carcinoma; Cirrhosis, Liver; Transmission Vertical
Keywords: Chronic hepatitis D; Hepatocellular Carcinoma; Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular; Hepatitis D, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 13 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Family Physicians: 1. 250 Family Physicians
- HDV Screening: 2. 20,000 HBsAg positive patients
  Interventions: Diagnostic Test: Anti Delta

INTERVENTIONS:
Diagnostic Test: Anti Delta — Anti Delta by ELISA
  Other Names: Fibroscan
  Groups: HDV Screening

SUMMARY:
The aim of these study to determine the prevalence of hepatitis Delta virus (HDV) infections and the prognosis of HDV patients in Turkey's southeast. The investigators intend to arrange training sessions for 250 family physicians in Diyarbakir, Batman, Mardin, and Sanliurfa in order to determine those goals. The investigators will talk about diagnosing hepatitis B virus (HBV), HDV, hepatitis C virus (HCV), and Human Immunodeficiency virus (HIV) infections during these events. To ensure that patients with simultaneous HDV infection are evaluated for HIV/HCV and to detect liver fibrosis with a non-invasive method.

DETAILED DESCRIPTION:
Study Objectives:

The aim of these study to determine the prevalence of HDV infections and the prognosis of HDV patients in Turkey's southeast. The investigators intend to arrange training sessions for 250 family physicians in Diyarbakir, Batman, Mardin, and Sanliurfa in order to determine those goals. The investigators will talk about diagnosing HBV, HDV, HCV, and HIV infections during these events. To ensure that patients with simultaneous HDV infection are evaluated for HIV/HCV and to detect liver fibrosis with a non-invasive method.

Primary Objectives:

To reveal the status of HDV infection in Turkey within the framework of the national hepatitis elimination program by providing training to family physicians.

Second Objectives:

* To determine the frequency and type of HDV in HBV patients (HDV/HCV co-infection).
* Providing HBV, HCV, HDV and HIV awareness training to family physicians.
* To determine the virological and liver fibrosis of patients with anti-Delta positivity.
* To determine the status of patients with HBV infection who are followed by family physicians.
* To ensure that patients with HDV infection are evaluated for liver cirrhosis and liver cancer.
* To determine the HDV/HIV co-infection rate.
* To determine the HDV/HCV co-infection rate.
* Determining the vertical transmission rate in viral hepatitis and contributing to elimination by emphasizing the importance of this rate.

Study Population:

To ensure that 20,000 patients with HBsAg positivity in Diyarbakir, Mardin, Batman and Sanliurfa are evaluated for HDV infection. To investigate HDV positive patients for liver fibrosis using the fibroscan method.

Number of Volunteers to Participate in the Study:

It is planned to include a total of 20,000 patients with HBsAg positivity from four provinces in this study.

Study Design:

Hepatitis Delta Virus infection poses a greater risk of developing both cirrhosis and liver cancer than other viral hepatitis agents. The Southeastern Anatolia region where HDV infection is most common in Turkey. It is planned to include four provinces (Diyarbakir, Batman, Mardin and Sanliurfa) in this study. In this study, family physicians will be reached through the Health Directorate of each province.

All Family Physicians will be educated about the prognosis and complications of HBV and especially HDV infection. The training will be carried out by the Infectious Diseases or Gastroenterology specialists of that province. Anti-Delta will be tested in all patients applying to health institutions. At the same time, all HBsAg positive patients followed by each family physician will be evaluated for the presence of HDV infection. All patients with anti-Delta positivity will be tested for HIV and HCV to determine their HDV/HIV co-infection and HDV/HCV co-infection status. Simultaneously, the liver fibrosis of patients with Anti-Delta positivity will be evaluated by the fibroscan method. Fibrosis-4 (FIB-4) and Child Pugh scoring will be performed on all patients simultaneously.

After receiving ethics committee approval for this study, the data collection process for family physicians' training and follow-up patients will be completed between April and July 2024. In total, it is anticipated to reach 250 Family Physicians in the entire region. In addition, demographic characteristics of HDV patients will be determined by reaching the Infectious Diseases and Gastroenterology Centers in four provinces. A five-question survey would be organized for all family physicians before and after the training in order to measure their knowledge level and evaluate the contribution of the training. This survey will be applied and analyzed via Slido.

After determining the biochemical and virological status of all HDV infections detected in four provinces, fibrosis of the liver will be measured with Fibroscan and FIB-4, which are non-invasive methods. As a result of the study, it is aimed to diagnose an estimated 1000 HDV-infected patients and score their liver fibrosis. It is aimed to complete the biochemical, virological, demographic and liver fibrosis status and statistical analyzes of all HDV-infected patients by 31.12.2024. The status of all patients in need of treatment or transplantation will be determined and their follow-up and treatment will be carried out in line with the recommendations of international and national treatment guidelines. The writing phase of all analyzed data will be completed and finalized by 31.01.2025.

One of the important reasons why both hepatitis B infection (HBV) and HDV infections are common is related to the fact that until recently vertical transmission was an important risk factor.

Both the diagnostic approach and follow-up and effective treatment options for HDV infections are still limited. It is also clearly known that HDV infection carries a higher risk of hepatocellular carcinoma (HCC) and cirrhosis than HBV infection. It is known that 90% of patients with viral hepatitis origin who are transplant candidates in our country have HDV infection.

ELIGIBILITY:
Inclusion Criteria:

* Adults (Age≥18)
* Being HBsAg positive for at least six months
* Being a citizen of the Republic of Türkiye

Exclusion Criteria:

* There are no exclusion criteria in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To ensure that 20,000 patients with HBsAg positivity in Diyarbakir, Mardin, Batman and Sanliurfa are evaluated for HDV infection. To investigate HDV positive patients for liver fibrosis using the fibroscan method.
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
The frequency of HDV in certain regions of Southern Anatolia | 01.04.2024-30.09.2024
  The primary endpoint of this study is to determine the frequency of HDV in certain regions of Southern Anatolia, and the virological and liver fibrosis status of patients with HDV infection.

SECONDARY OUTCOMES:
The rate of HIV and HCV co-infection in HDV positive patients | 01.04.2024-30.09.2024
  To determine the rate of HIV and HCV co-infection in HDV positive patients and to determine the demographic characteristics of HDV infected cases.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Kemal Çelen, MD, Principal Investigator — Dicle University, Medical Faculty, Department of Infectious Diseases
Locations (2):
- Turkey (Türkiye) (2):
  - Guven Hospital, Ankara
  - Dicle University, Faculty of Medicine, Diyarbakır

IPD SHARING:
Plan to Share IPD: No
Study data will be shared with researchers periodically.